CLINICAL TRIAL: NCT00635310
Title: Safety Profiles of Percutaneous Liver Biopsy in Hemodialysis Patients With Chronic Hepatitis C Pre-treated With 1-Deamino-8- D-Arginine Vasopressin
Brief Title: Safety Profiles of Liver Biopsy in Hemodialysis Patients With Chronic Viral Hepatitis Pre-treated With Vasopressin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 940211
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Hepatitis C; Chronic Hepatitis B; Biopsy; Hemodialysis
Keywords: Chronic hepatitis C; Chronic hepatitis B; Liver biopsy; Hemodialysis; 1-Deamino-8- D-Arginine Vasopressin
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HD patients with CHC or CHB (Active Comparator): Chronic hepatitis C (CHC) or chronic hepatitis B (CHB) patients with hemodialysis (HD), pretreated with DDAVP 0.3 ug/kg body weight infusion 30-60 minutes before percutaneous liver biopsies (PLBs)
  Interventions: Procedure: Percutaneous liver biopsy
- Ordinary patients with CHC or CHB (Active Comparator): Chronic hepatitis C (CHC) or chronic hepatitis B (CHB) patients with normal renal function (NRF) receiving percutaneous liver biopsies (PLBs)
  Interventions: Procedure: Percutaneous liver biopsy

INTERVENTIONS:
Procedure: Percutaneous liver biopsy — Two passes of PLB from the right hepatic lobe by US guidance (ToshibaTM PLF-308P, Toshiba Co. Ltd., Tokyo, Japan) and 16-gauge automatic cutting needles (Temno EvolutionTM, Allegiance, McGaw Park, IL, USA)
  Arms: HD patients with CHC or CHB
Procedure: Percutaneous liver biopsy — Two passes of PLB from the right hepatic lobe by US guidance (ToshibaTM PLF-308P, Toshiba Co. Ltd., Tokyo, Japan) and 16-gauge automatic cutting needles (Temno EvolutionTM, Allegiance, McGaw Park, IL, USA)
  Arms: Ordinary patients with CHC or CHB

SUMMARY:
Percutaneous liver biopsy (PLB) is the gold standard for grading necroinflammation and staging fibrosis in patients with chronic viral hepatitis. Whether the use of 1-deamino-8-D-arginine vasopressin (DDAVP) before PLBs in hemodialysis (HD) patients with chronic viral hepatitis has comparable safety profiles to those with normal renal function (NRF) has not been evaluated in prospective studies.

DETAILED DESCRIPTION:
Chronic viral hepatitis is common in dialysis patients, with the reported prevalence and annual incidence of 3-80% and 2.9%, respectively. Currently, percutaneous liver biopsy (PLB) remains the gold standard for grading necroinflammation and staging fibrosis in patients with liver diseases. In addition, liver histology can help clinicians determine the eligibility of renal transplantation, prognosis, and necessity of antiviral therapy in dialysis patients with chronic viral hepatitis. In chronic hepatitis patients with normal renal function (NRF), the risks of fatal and non-fatal hemorrhage after liver biopsies for non-malignant diseases were 0.04% and 0.16%, respectively. However, the relative risks of post-biopsy hemorrhage in CHC patients with end-stage renal disease to those with NRF remain disputed.

Deamino-8-D-arginine vasopressin (DDAVP), a synthetic analogue of vasopressin, is a commonly used hemostatic agent to treat uremic bleeding by inducing the release of von Willebrand factor (vWF) and factor VIII from their storage sites in endothelial cells.Previous studies have shown that one dose of 0.3-0.4μg/kg body weight DDAVP infusion for dialysis patients could normalize bleeding time (BT), and prevent surgical and renal biopsy bleeding. Nevertheless, two recent studies showed divergent liver biopsy-related bleeding complication rates (0% and 6%, respectively) in dialysis CHC patients pre-treated with DDAVP. Since most studies evaluating the safety of PLB in CHC patients with dialysis were small and retrospective in nature, and not controlled by the biopsy route, the type of biopsy needle, the use of ultrasound guidance, or the number of passes,further studies are urgently needed to solve this important issue. Thus, we aimed to conducted a large clinical trial to compare the safety profiles of PLB between CHC patients with hemodialysis (HD) who were pretreated with DDAVP and those with NRF by the same biopsy technique.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C (presence of anti-HCV and serum HCV RNA > 6 months)
* Chronic hepatitis B (presence of HBsAg > 6 months)
* Receiving regular hemodialysis or normal renal function (Creatinine < 1.5 x ULN)
* Receiving percutaneous liver biopsy (PLB)

Exclusion Criteria:

* Human immunodeficiency virus (HIV) co-infection
* Unwilling or contraindicated to receive percutaneous liver biopsy (PLB)
* Receiving liver biopsy without ultrasound (US) guidance or automatic cutting needles
* Did not receive 2 passes of liver biopsy
* Inadequate record of post-biopsy complications

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3520 (Estimated)
Dates: Start 2005-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Biopsy-related serious hemorrhage rate by intention-to-treat (ITT) analysis | 14 days

SECONDARY OUTCOMES:
Biopsy-related serious hemorrhage rate by per-protocol (PP) analysis | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital; Jia-Horng Kao, MD, Principal Investigator — National Taiwan University Hospital; Chun-Jen Liu, MD, Principal Investigator — National Taiwan University Hospital; Ming-Yang Lai, MD, Principal Investigator — National Taiwan University Hospital; Pei-Jer Chen, MD, Principal Investigator — National Taiwan University Hospital; Ding-Shinn Chen, MD, Principal Investigator — National Taiwan University Hospital; Cheng-Chao Liang, MD, Principal Investigator — Far Eastern Memorial Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Jou-Wei Lin, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Shih-I Chen, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Hung-Bin Tsai, MD, Principal Investigator — St. Martin De Porres Hospital; Peir-Haur Hung, MD, Principal Investigator — Chiayi Christian Hospital; Jun-Herng Chen, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (5):
- Taiwan (5):
  - Chiayi Christian Hospital, Chiayi City
  - St. Martin De Porres Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei